CLINICAL TRIAL: NCT03751215
Title: Anterior Chamber Depth (ACD) Variability Between the Clareon and Acrysof IOL: a Randomised Trial
Brief Title: Anterior Chamber Depth Variability Between Two Lenses With Different Materials
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clareon
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; Intraocular lens
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monofocal IOL (Experimental): Patients will be implanted with two different monofocal lenses (Clareon and AcrySof) during cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — During cataract surgery the patient is implanted with the monofocal IOL Clareon in one eye and the monofocal IOL AcrySof in the contralateral eye

SUMMARY:
Compare the change of the Anterior chamber depth (ACD) variability between the Clareon and the AcrySof Intraocular lens (IOL) after implantation over 6 months.

DETAILED DESCRIPTION:
Patients undergoing cataract surgery are often otherwise healthy and active with their only restriction being reduced visual quality. Within the past few years, intraocular lenses (IOLs) have been improved to fulfill the needs of these patients. Nowadays efforts are aiming for the enhancement of the patient vision and his subjective satisfaction postoperative.

One of the best ways to accomplish this is to have a perfect intraocular lens (IOL) power calculation. However, the best calculation can't help if the implanted intraocular lens (IOL) changes its position after implantation.

It should be considered that an anterior chamber depth (ACD) shift, decentration, tilt or rotation of an IOL could result in a reduction in visual quality. For an aspherical IOL, for instance, it is essential not to be decentrated and tilted more than 0.4 mm 2 (0.8 mm 3) and 7° 2 (10° 3), respectively. Otherwise it will be outperformed by a spherical IOL. The estimation of the post-operative intraocular lens (IOL) position and therefore the estimated anterior chamber depth (ACD) is presently the main source of error (35% 4 to 42% 5) in IOL power calculation and therefore for the refractive outcome of the patients after cataract surgery. Presently the pre-operatively measured ACD is taken into account for several IOL power calculation formulas, such as the Haigis formula, the Holladay II formula and the Olsen formula.

To manage a better outcome an IOL with less postoperative influence of the anterior chamber depth (ACD) is very important. To accomplish a smaller deviation after the operation of the anterior chamber depth (ACD) the haptic and the material of the lens is very important. The change of the anterior chamber depth (ACD) after cataract surgery can be easily measured by instruments like the IOL-Master 700, AC-Master and Lenstar. It must be considered that every person is different and that change of the anterior chamber depth (ACD) in different eyes can cause high measurement errors. The changes in two eyes of the same patient help to minimize the error. These can help to achieve a better outcome for future patients.

The hydrophobic acrylate of the Acrysof IOL has been modified to the new material in the Clareon IOL. This study will evaluate whether the new Clareon has non-inferior axial stability to the Acrysof.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract in both eyes
* Scheduled for bilateral cataract surgery
* Age 21 and older
* Written informed consent prior to recruitment
* Visual Acuity > 0.05

Exclusion Criteria:

* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)
* Any ophthalmic abnormality that could compromise visual function or the measurements
* Presence of potential zonular weakness such as pseudoexfoliation Syndrome, history of ocular trauma, previous ocular surgery.

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Anterior chamber depth (ACD) | 12 months
  The change in anterior chamber depth (ACD) before and after cataract surgery will be measured using the IOL Master 700 and compared between the two different IOLs.

SECONDARY OUTCOMES:
Distance visual acuity | 12 months
  Uncorrected and corrected distance visual acuity will be determined using ETDRS-charts in a distance of 4 metres and differences in refraction will be compared between the two IOLs.

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ullrich M, Ruiss M, Hienert J, Pilwachs C, Fisus AD, Georgiev S, Hirnschall N, Findl O. Anterior chamber depth variability between 2 hydrophobic acrylic 1-piece intraocular lenses: randomized trial. J Cataract Refract Surg. 2021 Nov 1;47(11):1460-1465. doi: 10.1097/j.jcrs.0000000000000668. PMID 33929807